CLINICAL TRIAL: NCT05000099
Title: Fighting Against Social Isolation in Times of Pandemic Corona Virus-19: the Role of Technology in Elderly Patients: The SILVER Study
Brief Title: the Role of Technology in Elderly Patients
Acronym: SILVER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Patrizia D'Amelio, associated professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2020-01125
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Anxiety; Depression; Aging; Social Isolation
MeSH Terms: conditions — Anxiety Disorders; Depression; Social Isolation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- phone calls: patients choosing phone calls as preferred communication technique
  Interventions: Other: video calls
- video call: patients choosing video calls as preferred communication technique
  Interventions: Other: video calls

INTERVENTIONS:
Other: video calls — A tablet for video-calls will be available for patients and families. Two video-calls of maximum 15' will be organized every week; in addition, patients will be allowed to do video-call upon request. Video-calls will be performed using Skype or WhatsApp video or Face-time
  Other Names: phone calls

SUMMARY:
Starting from December 2019, the Severe Acute Respiratory Syndrome Corona Virus-2 (SARS-COV-2) disease spread rapidly from China into the world, with about two Mio cases confirmed around the world. In Switzerland, more than 26'000 cases have been confirmed so far, and health authorities declared in March the needs for social isolation and have banned visits to hospitalized patients and to nursing home residents. Loneliness and isolation is a significant concern for the elderly patients as well as for their families that may significantly affect physical and mental health in both.

SILVER aims to evaluate the role of programmed video calls with families:

* on mood, anxiety, fear of death and pain perception in patients hospitalized or in nursing homes during the SARS-COV-2 pandemic.
* in relieving the familiar caregiver anxiety and fear of death of others
* in relieving the professional caregiver anxiety.

SILVER is an international study involving both acute, rehabilitation geriatric units and nursing homes; we will enroll all the patients present in the participating centers. Patients will be allowed to chose between video and phone calls, the following dimensions will be evaluated:

* Delirium risk: using the Confusion Assessment Method (CAM)
* Mood: using the 5-item Geriatric Depression Scale (GDS)
* Anxiety: using the Clinical Anxiety Scale (GAS).
* Fear of death (self and others): using the Collett-Lester scale. In parallel, health professionals and family caregivers will be evaluated for anxiety at baseline and every week after intervention set-up by the Clinical Anxiety Scale (CAS). Family caregivers will also be evaluated with the fear of death scale (sub-scale fear of death of others).

Finally, to evaluate the appreciation for video call communication in patients and caregivers we will use a Likert scale.

DETAILED DESCRIPTION:
Aims.

* To evaluate the role of video calls with families on mood, anxiety, fear of death and pain perception in patients hospitalized or in nursing homes during the SARS-CoV-2 pandemic.
* To evaluate the role of video calls in relieving family caregivers' anxiety and fear of death of their loved one.
* To evaluate the role of video calls in relieving health professionals' anxiety.

Methods. In order to reduce social isolation from their relatives and friends patients will be helped in joining them through video-calls thanks to the use of dedicated tablets and to the assistance provided by nurses, assistant-nurses, occupational therapists or neuropsychologists.

Population selection. All the patients in the participating centers fulfilling inclusion/exclusion criteria will be enrolled in SILVER.

Patients will be asked to chose between video and phone call, phone call will be allowed without any restriction to both video and usual care groups.

standardization of video calls: Two video-calls of maximum 15' will be administered every week; in addition, patients will be allowed to do video-call upon request. Video-calls will be performed using Skype or WhatsApp video or Face-time, the use of others app will be evaluated upon family's request.

Data collection for primary and secondary outcomes. Patients will be evaluated at baseline and every week with standardized scales to assess their mood, anxiety and delirium symptoms.

At baseline and at the end of the intervention we will evaluate the overall appreciation of the video call by the patients, their family caregiver, and the health professionals using a Likert scale and Anxiety: using the Geriatric Anxiety Scale (GAS).

In order to clarify the role of social connection through video calls on the patients' health, we will evaluate at baseline and after one week :

* Mood: using the 5-items Geriatric Depression Scale (GDS-5)
* Fear of death (self and others): using the Collett-Lester scale
* Delirium risk: using the Confusion Assessment Method (CAM) will be evaluated every day and will be analyzed ad day of delirium weekly.

In addition, the effect of video calls in professionals and in family caregivers will be evaluated as follows:

family and professional caregivers will be evaluated for anxiety at baseline and the end of intervention set-up by the Clinical anxiety (CAS). Familiar care-givers will also be evaluated with the fear of death scale (sub-scale fear of death of others) at the baseline and after one week.

Collection of other data.

In order to correct the statistical analyses for possible confounding variables the following data will be collected:

Age, gender, years of school, duration of hospitalization , type of hospital discharge, Mini Mental State Examination (MMSE), Clinical Dementia Rating (CDR) scale, Cumulative Illness Rating Scale (CIRS) index, Activity of Daily Living (ADL), Instrumental Activities of Daily Living (IADL).

ELIGIBILITY:
Inclusion Criteria:

* patients of 65 years and older hospitalized in the participating unit during the absence of visits due to the SARS-CoV2 pandemic.
* Patients and families willing to participate.

Exclusion Criteria:

* patients or families who refuse to participate.
* Clinical Dementia Rating (CDR) equal or higher than two.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: SILVER is an observational multicentre study. Patients hospitalized in two geriatric Unit in Switzerland (the Centre Hospitalier Universitaire Vaudois (CHUV) in Lausanne and the Hôpitaux Universitaire Genève (HUG) in Geneva,) and in one geriatric unit in Italy (Santa Misericordia Hospital in Perugia) and their families
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
4-point likert scale (LKRT) | 0-7 days
  appreciation of video calls by patients and families rage 0-4, 4 represent the better outcome
Geriatric anxiety scale (GAS-10) | 0-7 days
  measure of anxiety, The GAS-10 form, contains a total of 10 items, the answers are yes or no and the possible scores range from 0 to 10, with a cut-off point for anxiety at 6. The higher the score, the greater the anxiety.
Collett Lester Fear of Death scale (CL-FOD) for self and others | 0-7 days
  fear of death scale of patients, The CL-FODS contains 28 items, with seven items on each of the four subscales: Fear of Death of Self, Dying of Self, Death of Others, and Dying of Others. It is answered on a 5-point Likert format anchored as follows: 1 (not) and 5 (very). The total score in each subscale could range from 7 to 35, with higher scores denoting higher anxiety from death or dying.
geriatric depression scale (GDS-5) | 0-7 days
  mood evaluation for patients. the GDS-5 contains 5 items, the total score range from 0 to 5, the clinical cut-off for suspicion of depression is 2

SECONDARY OUTCOMES:
Collett Lester Fear of Death scale (CL-FOD) for others | 0-7 days
  fear of death scale of others for family

CONTACTS AND LOCATIONS:
Locations (1):
- Patrizia D'amelio, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durst AV, Graf CE, Ruggiero C, Zekry D, Boccardi V, Monney L, Joss I, Vuilloud K, Vespignani G, Bosshard W, Mecocci P, Bula CJ, D'Amelio P. Fighting social isolation in times of pandemic COVID-19: the role of video calls for older hospitalized patients. Aging Clin Exp Res. 2022 Sep;34(9):2245-2253. doi: 10.1007/s40520-022-02188-8. Epub 2022 Jul 6. PMID 35794314